CLINICAL TRIAL: NCT02062957
Title: Endovascular Function in Patients With Atrial Fibrillation
Brief Title: Endovascular Function in Atrial Fibrillation (AF) Patients
Acronym: HEAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guangzhen Zhong, associate professor, Beijing Chao Yang Hospital
Other Study IDs: NF81300148
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: PAT Result

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. recruit 50 patients with atrial fibrillation and 30 controls
2. endovascular function assessment with Peripheral Arterial Tonometry (PAT)
3. follow up the occurence of AF

ELIGIBILITY:
Inclusion Criteria:

* ≥2 paroxysmal (electrocardiographic documentation of at least 1) AF episodes lasting ≥1 hour in duration: (that terminate spontaneously within 7 days or cardioversion is performed within 48h of AF onset): or
* electrocardiographic documentation of 1 persistent AF episode: (sustained for ≥7 days or cardioversion is performed more than 48h after AF onset): or
* electrocardiographic documentation of 1 longstanding persistent AF episode: (continuous AF of duration >1 year).

Exclusion Criteria:

* patients with cerebralvascular disease
* patients with coronary disease
* patients with peripheric artery disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with AF
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
endovascular function results | Up to 24 weeks.
  The method to assess the endovascular function is PAT. The index is Reactive hyperemia index (RHI). RHI between patients and control will be compared.

SECONDARY OUTCOMES:
predictive effect of endovascular function on recurrence of AF | Up to 1 year
  We will do the multi-logistic analysis of the recurrence of AF.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Beijing, China